CLINICAL TRIAL: NCT00271180
Title: Medtronic CRDM Product Performance Report
Brief Title: Product Performance Report: Evaluate Long-term Reliability & Performance of Medtronic Marketed Cardiac Therapy Products
Acronym: PPR
Status: Recruiting | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 602
Record Dates: First submitted 2005-12-28; First posted 2005-12-30 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Arrhythmia; Bradycardia; Heart Failure; Sinus Tachycardia
Keywords: Cardiac Pacing; Implantable Cardioverter Defibrillator; pacemaker; Sinus Bradycardia
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia; Heart Failure; Tachycardia, Sinus | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Device

SUMMARY:
The main purpose of the Product Performance Report (formerly referred to as System Longevity Study) is to evaluate long-term performance of Medtronic market-released cardiac rhythm products by analyzing product survival probabilities.

DETAILED DESCRIPTION:
All Medtronic market-released leads and all market-released IPG, ICD and CRT devices are eligible to be included in this study.

ELIGIBILITY:
Subjects who meet the following inclusion criteria and do not meet any of the following exclusion criteria are eligible for enrollment.

Inclusion Criteria:

• Subject or appropriate legal guardians provide written informed consent and/or authorization for access to and use of health information as required by an institution's IRB/MEC/REB

AND one of the following must also apply:

* Subject is indicated for implant or within 30 days post-implant of at least one Medtronic market-released product used for a pacing, sensing or defibrillation application
* Subjects who participated in a qualifying study (IDE) of a Medtronic market-released product with complete implant and follow-up data and subject or appropriate legal guardian authorizes release of subject study data

Exclusion Criteria:

* Subjects who are, or will be inaccessible for follow-up
* Subjects with exclusion criteria required by local law (EMEA only)
* Subjects receiving an implant of a Medtronic device at a non-participating center and the implant data and current status cannot be confirmed within 30 days after implant
* Subjects implanted with a Medtronic device whose predetermined enrollment limit for that specific product has been exceeded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects implanted with Medtronic qualifying cardiac rhythm product.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 1983-01 (Actual); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Lead related complications for each lead model. | Ongoing: Implant to the cardiac lead is terminated from the study if the patient exit, patient death, or out-of-service (e.g. deactivated/inactive).
  All follow-up visits will be utilized in the analyses. This is an observational study that does not have a statistically powered primary hypothesis. Therefore, a specific study sample size is not applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Product Performance Report Study Leader, Study Chair — Medtronic
Locations (318):
- United States (112):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Chandler, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Bakersfield, California
  - Chula Vista, California
  - La Jolla, California
  - Los Angeles, California
  - Palm Springs, California
  - Rancho Mirage, California
  - Redwood City, California
  - Salinas, California
  - San Diego, California
  - Stanford, California
  - Torrance, California
  - Van Nuys, California
  - Ventura, California
  - Aurora, Colorado
  - Centennial, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Lakewood, Colorado
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Clearwater, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Panama City, Florida
  - Safety Harbor, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Evansville, Indiana
  - Indianapolis, Indiana
  - West Des Moines, Iowa
  - Kansas City, Kansas
  - Edgewood, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Clinton, Maryland
  - Hyattsville, Maryland
  - Salisbury, Maryland
  - Silver Spring, Maryland
  - Takoma Park, Maryland
  - Boston, Massachusetts
  - Lansing, Michigan
  - Marquette, Michigan
  - Ypsilanti, Michigan
  - Coon Rapids, Minnesota
  - Minneapolis, Minnesota
  - Robbinsdale, Minnesota
  - Rochester, Minnesota
  - Saint Cloud, Minnesota
  - Saint Paul, Minnesota
  - Hattiesburg, Mississippi
  - Columbia, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Eatontown, New Jersey
  - Marlton, New Jersey
  - Morristown, New Jersey
  - New Brunswick, New Jersey
  - Ocean City, New Jersey
  - Ridgewood, New Jersey
  - Albuquerque, New Mexico
  - Huntington, New York
  - Manhasset, New York
  - New York, New York
  - Poughkeepsie, New York
  - Utica, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Bethlehem, Pennsylvania
  - Danville, Pennsylvania
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Columbia, South Carolina
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Plano, Texas
  - The Woodlands, Texas
  - Tyler, Texas
  - Burlington, Vermont
  - Charlottesville, Virginia
  - Falls Church, Virginia
  - Olympia, Washington
  - Spokane, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Australia (4):
  - Chermside
  - Douglas
  - Murdoch
  - Southport
- Austria (4):
  - Graz
  - Innsbruck
  - Linz
  - Vienna
- Belgium (6):
  - Bruges
  - Brussels
  - Edegem
  - Leuven
  - Liège
  - Yvoir
- Canada (4):
  - Calgary
  - Kingston
  - Montreal
  - Québec
- China (14):
  - Beijing
  - Changsha
  - Dalian
  - Fuzhou
  - Guangzhou
  - Hangzhou
  - Harbin
  - Kunming
  - Nanchang
  - Shanghai
  - Shantou
  - Suzhou
  - Taiyuan
  - Tianjin
- Prague, Czechia
- Denmark (5):
  - Aarhus
  - Copenhagen
  - Hellerup
  - Hillerød
  - Odense
- Helsinki, Finland
- France (22):
  - Avignon
  - Bayonne
  - Brest
  - Caen
  - Chambray-lès-Tours
  - Clermont-Ferrand
  - Dijon
  - La Rochelle
  - La Tronche
  - Lille
  - Montpellier
  - Nantes
  - Neuilly-sur-Seine
  - Paris
  - Pessac
  - Pringy
  - Rennes
  - Saint-Priest-en-Jarez
  - Strasbourg
  - Toulouse
  - Vandœuvre-lès-Nancy
  - Villeurbanne
- Germany (17):
  - Aachen
  - Bad Oeynhausen
  - Bremen
  - Cologne
  - Dresden
  - Düsseldorf
  - Essen
  - Hamburg
  - Hanover
  - Heidelberg
  - Homburg
  - Jena
  - München
  - Münster
  - Tübingen
  - Ulm
  - Villingen-Schwenningen
- Greece (3):
  - Athens
  - Marousi
  - Thessaloniki
- Hong Kong, Hong Kong
- Budapest, Hungary
- Reykjavik, Iceland
- India (5):
  - Bangalore
  - Gūrgaon
  - Jaipur
  - Kochi
  - New Delhi
- Israel (4):
  - Ashkelon
  - Beersheba
  - Jerusalem
  - Ramat Gan
- Italy (12):
  - Ancona
  - Bari
  - Bologna
  - Brescia
  - Castrovillari
  - Cotignola
  - Lecce
  - Milan
  - Monza
  - Pisa
  - Taranto
  - Udine
- Japan (27):
  - Ageo
  - Bunkyō City
  - Gifu
  - Hidaka
  - Hiroshima
  - Kagoshima
  - Kamakura
  - Kawasaki
  - Kitakyushu
  - Koshigaya
  - Kumamoto
  - Kyoto
  - Mitaka
  - Nagoya
  - Niigata
  - Okayama
  - Ōsaka-sayama
  - Sapporo
  - Shinagawa-Ku
  - Shizuoka
  - Suita
  - Tokyo
  - Toyoake
  - Tsukuba
  - Urasoe
  - Yamagata
  - Yokohama
- Kuwait (2):
  - Hadiya
  - Kuwait City
- Kuala Lumpur, Malaysia
- Netherlands (10):
  - Amsterdam
  - Breda
  - Eindhoven
  - Enschede
  - Groningen
  - Leiden
  - Maastricht
  - Nieuwegein
  - Rotterdam
  - The Hague
- Christchurch, New Zealand
- Norway (3):
  - Bergen
  - Oslo
  - Trondheim
- Poland (3):
  - Poznan
  - Warsaw
  - Zabrze
- Portugal (5):
  - Carnaxide
  - Creixomil
  - Lisbon
  - Porto
  - Santarém
- Saudi Arabia (2):
  - Jeddah
  - Riyadh
- Belgrade, Serbia
- Slovakia (2):
  - Bratislava
  - Košice
- Ljubljana, Slovenia
- South Korea (5):
  - Cheongju-si
  - Daejeon
  - Gyeonggi-do
  - Seoul
  - Suwon
- Spain (14):
  - A Coruña
  - Barcelona
  - Córdoba
  - Girona
  - Granada
  - Madrid
  - Palma de Mallorca
  - Salamanca
  - Santa Cruz de Tenerife
  - Santiago de Compostela
  - Toledo
  - Valencia
  - Valladolid
  - Vitoria-Gasteiz
- Sweden (4):
  - Gothenburg
  - Lund
  - Skövde
  - Uppsala
- Switzerland (7):
  - Basel
  - Bern
  - Fribourg
  - Geneva
  - Lausanne
  - Lugano
  - Zurich
- United Kingdom (13):
  - Birmingham
  - Blackpool
  - Bristol
  - Leeds
  - Leicester
  - Liverpool
  - London
  - Manchester
  - Middlesbrough
  - Northampton
  - Nottingham
  - Sheffield
  - Southampton